CLINICAL TRIAL: NCT06608485
Title: A Prospective, Single-Arm Multi-Center Study of the HARMONIC™ 700, 5 mm Diameter Shears With Advanced Hemostasis in Pediatric Surgical Procedures (General) and Adult Surgical Procedures (General, Gynecological, Urological, and Thoracic)
Brief Title: A Study of HARMONIC 700 Shears With Advanced Hemostasis in Pediatric and Adult Surgical Procedures
Status: Recruiting | Type: Observational
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: ENG202301; ENG202301 (Other: Ethicon Endo Surgery)
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Surgical Procedures; Adult Surgical Procedures; Adult Gynecological Procedures; Adult Urological Procedures; Adult Thoracic Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Pediatric; Adult Surgical Procedures (HARMONIC 700 Shears): This prospective study will involve collection of clinical data in a post-market setting from pediatric surgical procedures (general) and adult surgical procedures (general, gynecological, urological, and thoracic surgical procedures). Investigators will perform each procedure using the device in compliance with their standard surgical approach and the HARMONIC 700 Shears instruction for use (IFU). All subjects enrolled will be followed post-operatively through discharge and again at approximately 28 days post-surgery.
  Interventions: Device: HARMONIC 700 Shears

INTERVENTIONS:
Device: HARMONIC 700 Shears — There is no intervention, beyond necessary clinical care, in this study. HARMONIC 700 Shears for vessel transection were used according to instructions for use.

SUMMARY:
The main purpose of this study is to demonstrate acceptable performance and assess safety of the HARMONIC 700 Shears device in a post-market setting when used per the instructions for use in pediatric and adult surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

Pediatric participants

* Non-emergent procedure (general) where at least one vessel is planned to be transected by the HARMONIC 700 Shears per the IFU
* Less than 18 years of age at the time of procedure
* Participant's parent/legal guardian must give permission to participate in the study and provide written informed consent for the participant Adult participants
* Elective procedure (general, gynecological, urological, or thoracic) where at least one vessel is planned to be transected by the HARMONIC 700 Shears per the IFU
* Elective procedure (general, gynecological, urological, or thoracic) where at least one vessel is planned to be transected by the HARMONIC 700 Shears per the IFU

Exclusion Criteria:

Preoperative

* Physical or psychological condition which would impair study participation
* Participants of childbearing potential who are pregnant
* Enrollment in a concurrent interventional clinical study that could impact the study endpoints Intraoperative
* HARMONIC 700 Shears were not attempted to be used for at least one single vessel transection during the surgical procedure

Max Age: 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include pediatric participants aged less than (<) 18 years of age and adult participants of at least 18 years of age in whom at least one vessel is planned to be transected by the HARMONIC 700 Shears as per the instructions for use (IFU).
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Number of Vessel Transections With an Achievement of Grade 3 or Lower Hemostasis | Intraoperative
  Number of vessel transection with achievement of Grade 3 or lower hemostasis for each vessel transection will be reported as per the grading scale as follows- Grade 1: no bleeding at transection site; Grade 2: minor bleeding at transection site, no intervention needed; Grade 3: minor bleeding at transection site, mild intervention needed, use of compression, basic energy devices (monopolar and/or bipolar) and/or touch-ups with HARMONIC 700 Shears; Grade 4: significant bleeding (for example [e.g.], pulsatile blood flow, venous pooling) requiring intervention such as extensive coagulation or ligation with use of additional hemostatic measures.
Number of Participants with Device-Related Adverse Events (AEs) | Up to approximately 1 year and 7 months
  An AE is defined as any untoward medical occurrence, regardless of its relationship to the study device or the study procedure. An untoward medical occurrence includes any new, undesirable medical experience or worsening of a pre-existing condition, which occurs throughout the duration of the clinical study.

SECONDARY OUTCOMES:
Number of Vessel Transections With an Achievement of Grade 3 or Lower Hemostasis for Each Vessel Transection of Diameter Greater Than (>) 5 to 7 Millimeter (mm) | Intraoperative
  Number of vessel transections with achievement of Grade 3 or lower hemostasis for each vessel transection of diameter > 5 to 7 mm will be reported as per the grading scale as follows- Grade 1: no bleeding at transection site; Grade 2: minor bleeding at transection site, no intervention needed; Grade 3: minor bleeding at transection site, mild intervention needed, use of compression, basic energy devices (monopolar and/or bipolar) and/or touch-ups with HARMONIC 700 Shears; Grade 4: significant bleeding (e.g., pulsatile blood flow, venous pooling) requiring intervention such as extensive coagulation or ligation with use of additional hemostatic measures.

CONTACTS AND LOCATIONS:
Overall Officials: Ethicon Endo-Surgery, Inc. Clinical Trial, Study Director — Ethicon Endo-Surgery, Inc.
Locations (8):
- United States (4):
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - NextStage Clinical Research, Wichita, Kansas
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - The Methodist Hospital Research Institute D B A Houston Methodist Research Institute, Houston, Texas
- Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec, Canada
- United Kingdom (3):
  - Dorset County Hospital Nhs Foundation Trust, Dorchester
  - Western General Hospital, Edinburgh
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No